CLINICAL TRIAL: NCT05583604
Title: Managed Access Programs for AIN457, Secukinumab
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457M2002M
Record Dates: First submitted 2022-10-04; First posted 2022-10-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: MAP; Manage Access Program; Hidradenitis suppurativa (HS); AIN457; secukinumab; Cosentyx
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — secukinumab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: secukinumab — Patients receive secukinumab
  Other Names: Cosentyx, AIN457

SUMMARY:
The purpose of this registration is to list Managed Access Programs (MAPs) related to AIN457, secukinumab

DETAILED DESCRIPTION:
CAIN457M2002M - Available - Managed Access Program (MAP) Cohort Treatment Plan CAIN457M2002M to provide access to Secukinumab for adult and adolescent patients with Hidradenitis Suppurativa (HS)

ELIGIBILITY:
Inclusion Criteria:

* An independent request should be received from a licensed physician (in some instances from Health Authorities, Institutions or Governments).
* The patient has a serious or life-threatening disease or condition and no comparable or satisfactory alternative therapy is available for diagnosis, monitoring or treatment; patient is not medically eligible for available treatment alternatives or has exhausted all available treatment options.
* The patient is not eligible or able to enroll in a Novartis clinical trial or continue participation in a Novartis clinical trial.
* There is a potential patient benefit to justify the potential risk of the treatment use, and the potential risk is not unreasonable in the context of the disease or condition to be treated.
* The patient must meet any other medical criteria established by the medical experts responsible for the product or by the Health Authority in a country (as applicable).
* Provision of the product will not interfere with the initiation, conduct or completion of a Novartis clinical trial or overall development program.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals